CLINICAL TRIAL: NCT00335166
Title: A Multicenter, Randomized, Double Blind, Parallel-Group Placebo and Pramipexole Controlled Study to Assess Efficacy and Safety of SLV308 Monotherapy in the Treatment of Patients With Early Stage Parkinson's Disease.
Brief Title: SLV 308 and Pramipexole for Treatment of Patients With Early Parkinson Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Solvay Pharmaceuticals (Industry)
Responsible Party: Ellen van Kleef, Solvay Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: S308.3.003; Not requested yet
Record Dates: First submitted 2006-06-08; First posted 2006-06-09 (Estimated); Last update posted 2008-04-03 (Estimated); Status verified 2008-04

CONDITIONS: Early Stage Parkinson Disease
Keywords: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Pramipexole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: Pardaprunox
- 2 (Active Comparator)
  Interventions: Drug: pramipexole
- 3 (Placebo Comparator)
  Interventions: Drug: Placebo Comparator

INTERVENTIONS:
Drug: Pardaprunox — 12-42 mg
  Arms: 1
Drug: pramipexole — 1.5-4.5 mg
  Arms: 2
Drug: Placebo Comparator — Placebo
  Arms: 3

SUMMARY:
This is a multicenter, randomized, double blind, parallel group study of 6 months' treatment with SLV308 as monotherapy in patients with early stage PD. An open label safety extension to this study is planned as a separate protocol for patients who are willing and eligible to participate.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic Parkinson's Disease, Modified Hoehn & Yahr up to stage III, UPDRS motor score (part III) must have a total of at least 10 at baseline.

Exclusion Criteria:

* Diagnosis is unclear or a suspicion of other parkinsonian syndromes,
* Patients who have undergone surgery for the treatment of PD,
* Current presence of dyskinesias,
* Motor fluctuations or loss of postural reflexes,
* A history of non-response to an adequate course of l-dopa or a dopamine agonist,
* Patients for whom previously treatment with dopamine agonists needed to terminate because of induction of psychosis (i.e. hallucinations) and /or sleep attacks.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2006-11; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
UPDRS part 3 (motor score)and change from baseline to 24 weeks maintenance treatment | 24 weeks

SECONDARY OUTCOMES:
UPDRS part 2 (ADL score); CGI-Improvement; PDQ-39 total score: all change from baseline to 24 weeks maintenance treatment. | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Director Solvay, Study Director — Solvay Pharmaceuticals
Locations (89):
- United States (17):
  - 419, Birmingham, Alabama
  - 413, Oceanside, California
  - 408, Oxnard, California
  - 422, New Haven, Connecticut
  - 403, Boca Raton, Florida
  - 411, Sarasota, Florida
  - 421, Augusta, Georgia
  - 410, Fort Wayne, Indiana
  - 417, Lexington, Kentucky
  - 405, Boston, Massachusetts
  - 420, Boston, Massachusetts
  - 415, Grand Rapids, Michigan
  - 416, Golden Valley, Minnesota
  - 406, Minneapolis, Minnesota
  - 418, Albany, New York
  - 424, Charlotte, North Carolina
  - 412, Raleigh, North Carolina
- Australia (4):
  - 303, Bedford Park
  - 304, Cheltenham
  - 301, Concord
  - 302, Westmead
- Czechia (6):
  - 315, Kralove
  - 313, Olomouc
  - 310, Ostrava
  - 314, Ostrava
  - 312, Pardubice
  - 311, Pilsen
- Estonia (2):
  - 320, Tallinn
  - 321, Tartu
- France (3):
  - 323, Aix-en-Provence
  - 324, Toulon
  - 325, Toulouse
- Germany (7):
  - 332, Bochum
  - 331, Göttingen
  - 329, Heidelberg
  - 327, Homburg
  - 330, Leipzig
  - 328, Lübeck
  - 326, Wiesbaden
- India (5):
  - 338, Bangalore
  - 339, Hyderabad
  - 337, Kerala
  - 336, Mumbai
  - 340, Mumbai
- Italy (6):
  - 347, Arcugnano (VI)
  - 348, Grosseto GR
  - 346, Lido Di Camaiore (LU)
  - 344, Pescara
  - 343, Roma
  - 345, Roma
- Lithuania (3):
  - 428, Kaunas
  - 427, Vilnius
  - 429, Vilnius
- Malaysia (3):
  - 355, Kelantan
  - 357, Kuala Lumpur
  - 356, Pulau Pinang
- Netherlands (5):
  - 361, 's-Hertogenbosch
  - 364, Eindhoven
  - 363, Emmen
  - 362, Groningen
  - 360, RM Groningen
- Poland (9):
  - 373, Gdansk
  - 371, Kalisz
  - 369, Katowice
  - 374, Katowice
  - 365, Krakow
  - 368, Leszno
  - 366, Lublin
  - 370, Mosina
  - 367, Torun
- Portugal (2):
  - 376, Coimbra
  - 375, Lisbon
- South Africa (5):
  - 377, Cape Town
  - 378, Cape Town
  - 380, Gauteng
  - 381, Pretoria
  - 379, Sandton
- Spain (3):
  - 383, Barcelona
  - 384, Colmenar Viejo
  - 382, Donostia / San Sebastian
- Taiwan (5):
  - 388, Hualien City
  - 387, Kaohsiung City
  - 389, Kaohsiung Hsien
  - 386, Kweishan
  - 385, Taipei
- Thailand (3):
  - 391, Bangkok
  - 393, Bangkok
  - 394, Ubonratchathani Province
- 396, Blackpool, United Kingdom

REFERENCES:
- [Derived] Sampaio C, Bronzova J, Hauser RA, Lang AE, Rascol O, van de Witte SV, Theeuwes AA; Rembrandt/Vermeer Study Groups. Pardoprunox in early Parkinson's disease: results from 2 large, randomized double-blind trials. Mov Disord. 2011 Jul;26(8):1464-76. doi: 10.1002/mds.23590. Epub 2011 May 3. PMID 21542016